CLINICAL TRIAL: NCT03905330
Title: MRX-502: Randomized Double-blind Placebo-controlled Phase 3 Study to Evaluate the Efficacy and Safety of Maralixibat in the Treatment of Subjects With Progressive Familial Intrahepatic Cholestasis (PFIC) - MARCH-PFIC
Brief Title: A Study to Evaluate the Efficacy and Safety of Maralixibat in Subjects With Progressive Familial Intrahepatic Cholestasis (MARCH-PFIC)
Acronym: MARCH-PFIC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mirum Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MRX-502; 2019-001211-22 (EudraCT Number)
Record Dates: First submitted 2019-04-01; First posted 2019-04-05 (Actual); Results first posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Progressive Familial Intrahepatic Cholestasis (PFIC)
Keywords: Cholestasis; Maralixibat; Mutation; PFIC; PFIC2; Bile Duct Diseases; Liver Diseases; Biliary Tract Diseases; Digestive System Diseases; Pediatric
MeSH Terms: conditions — Cholestasis, progressive familial intrahepatic 1; Cholestasis; Bile Duct Diseases; Liver Diseases; Biliary Tract Diseases; Digestive System Diseases | interventions — maralixibat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Maralixibat (Experimental): Participants will receive Maralixibat oral solution (up to 600 microgram per kilogram [mcg/kg]) orally twice daily for 26 weeks.
  Interventions: Drug: Maralixibat
- Placebo (Placebo Comparator): Participants will receive placebo matched to maralixibat oral solution twice daily for 26 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Maralixibat — Maralixibat oral solution (up to 600 mcg/kg) orally twice daily for 26 weeks.
  Other Names: Formerly LUM001 and SHP625
  Arms: Maralixibat
Other: Placebo — Placebo matching to maralixibat orally twice daily for 26 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether the investigational treatment (maralixibat) is safe and effective in pediatric participants with Progressive Familial Intrahepatic Cholestasis (PFIC).

DETAILED DESCRIPTION:
This study was conducted at multiple sites in North America, Europe, Asia and South America.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent and assent (as applicable) per Institutional Review Board/Ethics Committee (IRB/EC)
2. Male or female subjects with a body weight ≥5 kg, who are ≥12 months and <18 years of age at time of baseline
3. Cholestasis as manifested by total sBA ≥3× ULN (applies to primary cohort only)
4. An average AM ItchRO(Obs) score ≥1.5 during 4 consecutive weeks of the screening period, leading to the baseline visit (Visit 1)
5. Completion of at least 21 valid* morning ItchRO(Obs) entries during 4 consecutive weeks of the screening period, leading to the baseline visit (Visit 1) (*valid = completed and not answered as "I don't know"; maximum allowed invalid reports = 7, no more than 2 invalid reports during the last 7 days before randomization)
6. Diagnosis of PFIC based on the following:

   * Chronic cholestasis as manifested by persistent (>6 months) pruritus in addition to biochemical abnormalities and/or pathological evidence of progressive liver disease and
   * Primary Cohort: Subjects with genetic testing results consistent with biallelic disease-causing variation in ABCB11 (PFIC2), based on standard of care genotyping
   * Supplemental Cohort: i. Subjects with genetic testing results consistent with biallelic disease-causing variation in ATP8B1 (PFIC1), ABCB4 (PFIC3), or TJP2 (PFIC4), based on standard of care genotyping. ii. Subjects with PFIC phenotype without a known mutation or with another known mutation not described above or with intermittent cholestasis as manifested by fluctuating sBA levels. iii. Subjects with PFIC after internal or external biliary diversion surgery or for whom internal or external biliary diversion surgery was reversed.
7. Male and females of non-childbearing potential. Males and non-pregnant, non-lactating females of childbearing potential who are sexually active must agree to use acceptable methods of contraception during the study and 30 days following the last dose of the study medication. Females of childbearing potential must have a negative pregnancy test
8. Access to email or phone for scheduled remote visits
9. Ability to read and understand the questionnaires (both caregivers and subjects above the age of assent)
10. Access to consistent caregiver(s) during the study
11. Subject and caregiver willingness to comply with all study visits and requirements.

Exclusion Criteria:

1. Predicted complete absence of bile salt excretion pump (BSEP) function based on the type of ABCB11 mutation (PFIC2), as determined by a standard of care genotyping (applies to primary cohort only). Subjects can enter the study in the Supplemental Cohort (under inclusion criteria 6.ii or 6.iii).
2. Recurrent intrahepatic cholestasis, indicated by a history of sBA levels <3x ULN or intermittent pruritus (applies to primary cohort only)
3. Current or recent history (<1 year) of atopic dermatitis or other non-cholestatic diseases associated with pruritus.
4. History of surgical disruption of the enterohepatic circulation (applies to primary cohort only)
5. Chronic diarrhea requiring intravenous fluid or nutritional intervention for the diarrhea and/or its sequelae at screening or during the 6 months prior to screening
6. Previous or need for imminent liver transplant
7. Decompensated cirrhosis (international normalized ratio [INR] >1.5, albumin <30 g/L, history or presence of clinically significant ascites, variceal hemorrhage, and/or encephalopathy)
8. ALT or total serum bilirubin (TSB) >15× ULN at screening
9. Presence of other liver disease
10. Presence of any other disease or condition known to interfere with the absorption, distribution, metabolism or excretion of drugs, including bile salt metabolism in the intestine (e.g., inflammatory bowel disease), per Investigator discretion
11. Possibly malignant liver mass on imaging, including screening ultrasound
12. Known diagnosis of human immunodeficiency virus (HIV) infection
13. Any prior cancer diagnosis (except for in situ carcinoma) within 5 years of the screening visit (Visit 0)
14. Any known history of alcohol or substance abuse
15. Administration of bile acids or lipid binding resins, or phenylbutyrates during the screening period
16. Criterion has been deleted as of Amendment 3
17. Administration of any investigational drug, biologic, or medical device during the screening period
18. Previous use of an ileal bile acid transporter inhibitor (IBATi)
19. History of non-adherence to medical regimens, unreliability, medical condition, mental instability or cognitive impairment that, in the opinion of the Investigator or Sponsor medical monitor, could compromise the validity of informed consent, compromise the safety of the subject, or lead to nonadherence with the study protocol or inability to conduct the study procedures
20. Known hypersensitivity to maralixibat or any of its excipients.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 93 (Actual)
Dates: Start 2019-07-09 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (31):
- United States (11):
  - Children's Hospital Los Angeles CHLA, Los Angeles, California
  - Medstar Georgetown University Hospital, Washington D.C., District of Columbia
  - Advent Health, Orlando, Florida
  - The Children's Hospital at Montefiore Yeshiva University - Montefiore Medical Center, New York, New York
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Cleveland Clinic - Pediatric Institute, Cleveland, Ohio
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas - UT Southwestern Medical Center, Dallas, Texas
  - University of Texas, Health Science Center San Antonio, San Antonio, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Hospital Italiano de Buenos Aires, Buenos Aires, Argentina
- Medizinische Universität Wien, Universitätsklinik für Kinder- und Jugendheilkunde, Vienna, Austria
- Universite Catholique de Louvain (UCLouvain) - Cliniques Universitaires Saint-Luc, Brussels, Belgium
- Sociedade Beneficente de Senhoras Hospital Sírio-Libanês, São Paulo, Brazil
- University of Alberta - Women and Children's Health Research Institute, Edmonton, Canada
- Fundacion Cardioinfantil - Departamento de Investigaciones, Bogotá, Colombia
- France (3):
  - Hospices Civils de Lyon - Hopital Femme Mere Enfant Service de Gastroenterologie, Hepatologie et Nutrition, Lyon
  - CHU de Marseille, Hôpital de la Timone, Marseille
  - CHU de Toulouse - Hôpital des Enfants, Toulouse
- Medizinische Hochschule Hannover, Hanover, Germany
- Semmelweis Egyetem - Altalanos Orvostudomanyi Kar (SE AOK), Budapest, Hungary
- Italy (2):
  - Hospital Papa Giovanni XXIII / Unità di Pediatria, Bergamo
  - Ospedale Pediatrico Bambino Gesu, Roma
- Hotel Dieu de France, Beirut, Lebanon
- Consultario de Joshue David Covarrubias Esquer, Zapopan, Mexico
- Instytut Pomnik Centrum Zdrowia Dziecka, Warsaw, Poland
- KK Women's and Children's Hospital, Singapore, Singapore
- Koc University Hospital, Istanbul, Turkey (Türkiye)
- United Kingdom (2):
  - Birmingham Children's Hospital, Birmingham
  - King's College Hospital NHS, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Miethke AG, Moukarzel A, Porta G, Covarrubias Esquer J, Czubkowski P, Ordonez F, Mosca A, Aqul AA, Squires RH, Sokal E, D'Agostino D, Baumann U, D'Antiga L, Kasi N, Laborde N, Arikan C, Lin CH, Gilmour S, Mittal N, Chiou FK, Horslen SP, Huber WD, Jaecklin T, Nunes T, Lascau A, Longpre L, Mogul DB, Garner W, Vig P, Hupertz VF, Gonzalez-Peralta RP, Ekong U, Hartley J, Laverdure N, Ovchinsky N, Thompson RJ. Maralixibat in progressive familial intrahepatic cholestasis (MARCH-PFIC): a multicentre, randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Gastroenterol Hepatol. 2024 Jul;9(7):620-631. doi: 10.1016/S2468-1253(24)00080-3. Epub 2024 May 6. PMID 38723644
- See also: Genetics Home Reference - PFIC — https://ghr.nlm.nih.gov/condition/progressive-familial-intrahepatic-cholestasis
- See also: US FDA Resources — https://clinicaltrials.gov/ct2/info/fdalinks
- See also: Mirum Pharmaceuticals homepage — https://mirumpharma.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 93 participants were enrolled at 29 sites in 16 countries (Argentina, Austria, Belgium, Brazil, Canada, Colombia, France, Germany, Italy, Lebanon, Mexico, Poland, Singapore, Turkey, United Kingdom, and United States).
Pre-assignment Details: The screening period starts when informed consent (or assent as applicable) is signed. The duration of the screening period is up to 6 weeks during which all procedures listed for the screening visit must be completed. A total of 125 patients were screened for the study. 32 of these patients were screen failures.
Groups:
- Maralixibat: Maralixibat up to 600 mcg/kg twice daily
- Placebo: Corresponding placebo
Period: Overall Study
Arm/Group | Maralixibat | Placebo
Started | 47 | 46
Dosed 150 ug/kg BID (150 ug/kg BID planned for 1 week) | 47 | 0
Dosed 300 ug/kg BID (300 ug/kg BID planned for 1 week) | 46 | 0
Dosed 450 ug/kg BID (450 ug/kg BID planned for 1 week) | 45 | 0
Dosed 600 ug/kg BID (600 ug/kg BID planned for 23 weeks) | 45 | 0
Completed | 44 | 42
Not Completed | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Maralixibat: After a screening period of up to 6 weeks, subjects were randomized 1:1 to receive either maralixibat or placebo. The Dose Escalation period (4-6 weeks) was followed by a stable dosing period (20-22 weeks) and a 7 days Safety Follow-up period for subjects discontinuing early and for subjects not enrolling into the extension Study MRX-503.
- Placebo: Participants received a corresponding placebo.
- Total: Total of all reporting groups
Arm/Group | Maralixibat | Placebo | Total
Number analyzed (Participants) | 47 | 46 | 93
Age, Categorical [Count of Participants; unit: Participants] — Population: The primary cohort and PFIC cohort are not mutually exclusive. Specifically, the primary cohort is fully contained in the PFIC cohort. The total population (n=93) consists of the primary cohort (n=31), the additional subjects in the PFIC cohort (n=33) and an additional 29 subjects for whom we did not run any primary or secondary efficacy analyses.
  Participants
    All subjects: <=18 years | 47 | 46 | 93
    All subjects: Between 18 and 65 years | 0 | 0 | 0
    All subjects: >=65 years | 0 | 0 | 0
    Primary Cohort: number analyzed (Participants) | 14 | 17 | 31
    Primary Cohort: <=18 years | 14 | 17 | 31
    Primary Cohort: Between 18 and 65 years | 0 | 0 | 0
    Primary Cohort: >=65 years | 0 | 0 | 0
    PFIC cohort: number analyzed (Participants) | 33 | 31 | 64
    PFIC cohort: <=18 years | 33 | 31 | 64
    PFIC cohort: Between 18 and 65 years | 0 | 0 | 0
    PFIC cohort: >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The primary cohort and PFIC cohort are not mutually exclusive. Specifically, the primary cohort is fully contained in the PFIC cohort. The total population (n=93) consists of the primary cohort (n=31), the additional subjects in the PFIC cohort (n=33) and an additional 29 subjects for whom we did not run any primary or secondary efficacy analyses.
  years
    All subjects | 4.8 (4.15) | 4.7 (3.57) | 4.7 (3.85)
    Primary Cohort: number analyzed (Participants) | 14 | 17 | 31
    Primary Cohort | 6.3 (5.24) | 4.2 (3.56) | 5.1 (4.45)
    PFIC Cohort: number analyzed (Participants) | 33 | 31 | 64
    PFIC Cohort | 4.9 (4.10) | 4.4 (3.61) | 4.6 (3.85)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The primary cohort and PFIC cohort are not mutually exclusive. Specifically, the primary cohort is fully contained in the PFIC cohort. The total population (n=93) consists of the primary cohort (n=31), the additional subjects in the PFIC cohort (n=33) and an additional 29 subjects for whom we did not run any primary or secondary efficacy analyses.
  Participants
    All subjects: Female | 27 | 24 | 51
    All subjects: Male | 20 | 22 | 42
    Primary Cohort: number analyzed (Participants) | 14 | 17 | 31
    Primary Cohort: Female | 7 | 11 | 18
    Primary Cohort: Male | 7 | 6 | 13
    PFIC Cohort: number analyzed (Participants) | 33 | 31 | 64
    PFIC Cohort: Female | 16 | 18 | 34
    PFIC Cohort: Male | 17 | 13 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The primary cohort and PFIC cohort are not mutually exclusive. Specifically, the primary cohort is fully contained in the PFIC cohort. The total population (n=93) consists of the primary cohort (n=31), the additional subjects in the PFIC cohort (n=33) and an additional 29 subjects for whom we did not run any primary or secondary efficacy analyses.
  Participants
    All subjects: Hispanic or Latino | 18 | 17 | 35
    All subjects: Not Hispanic or Latino | 28 | 27 | 55
    All subjects: Unknown or Not Reported | 1 | 2 | 3
    Primary Cohort: number analyzed (Participants) | 14 | 17 | 31
    Primary Cohort: Hispanic or Latino | 9 | 7 | 16
    Primary Cohort: Not Hispanic or Latino | 5 | 9 | 14
    Primary Cohort: Unknown or Not Reported | 0 | 1 | 1
    PFIC Cohort: number analyzed (Participants) | 33 | 31 | 64
    PFIC Cohort: Hispanic or Latino | 16 | 13 | 29
    PFIC Cohort: Not Hispanic or Latino | 17 | 16 | 33
    PFIC Cohort: Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The primary cohort and PFIC cohort are not mutually exclusive. Specifically, the primary cohort is fully contained in the PFIC cohort. The total population (n=93) consists of the primary cohort (n=31), the additional subjects in the PFIC cohort (n=33) and an additional 29 subjects for whom we did not run any primary or secondary efficacy analyses.
  Participants
    All subjects: American Indian or Alaska Native | 3 | 4 | 7
    All subjects: Asian | 3 | 0 | 3
    All subjects: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    All subjects: Black or African American | 1 | 2 | 3
    All subjects: White | 36 | 34 | 70
    All subjects: More than one race | 3 | 4 | 7
    All subjects: Unknown or Not Reported | 1 | 2 | 3
    Primary Cohort: number analyzed (Participants) | 14 | 17 | 31
    Primary Cohort: American Indian or Alaska Native | 3 | 3 | 6
    Primary Cohort: Asian | 0 | 0 | 0
    Primary Cohort: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Primary Cohort: Black or African American | 1 | 2 | 3
    Primary Cohort: White | 9 | 9 | 18
    Primary Cohort: More than one race | 1 | 2 | 3
    Primary Cohort: Unknown or Not Reported | 0 | 1 | 1
    PFIC Cohort: number analyzed (Participants) | 33 | 31 | 64
    PFIC Cohort: American Indian or Alaska Native | 3 | 4 | 7
    PFIC Cohort: Asian | 3 | 0 | 3
    PFIC Cohort: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    PFIC Cohort: Black or African American | 1 | 2 | 3
    PFIC Cohort: White | 24 | 19 | 43
    PFIC Cohort: More than one race | 2 | 4 | 6
    PFIC Cohort: Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants] — Measure Analysis Population Description: The primary cohort and PFIC cohort are not mutually exclusive. Specifically, the primary cohort is fully contained in the PFIC cohort. The total population (n=93) consists of the primary cohort (n=31), the additional subjects in the PFIC cohort (n=33) and an additional 29 subjects for whom we did not run any primary or secondary efficacy analyses.
  participants
    Argentina | 2 | 1 | 3
    Austria | 1 | 1 | 2
    Belgium | 3 | 0 | 3
    Brazil | 7 | 3 | 10
    Canada | 1 | 1 | 2
    Colombia | 2 | 4 | 6
    France | 1 | 2 | 3
    Germany | 1 | 1 | 2
    Italy | 2 | 4 | 6
    Lebanon | 6 | 8 | 14
    Mexico | 3 | 5 | 8
    Poland | 4 | 2 | 6
    Singapore | 2 | 0 | 2
    Turkey | 1 | 1 | 2
    United Kingdom | 2 | 0 | 2
    United States | 9 | 13 | 22

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in the Average Morning ItchRO(Obs) Severity Score in the Primary Cohort
Description: The primary efficacy endpoint is the mean change in the average morning ItchRO(Obs) severity score between baseline and Weeks 15-26, using 4-week average morning ItchRO(Obs) severity scores (Mixed Model Repeated Measures). The baseline average morning ItchRO(Obs) severity score is defined as the 4-week average morning ItchRO(Obs) severity score prior to the first dose of the study medication.
  ItchRo(Obs) Severity Score = Itch Reported Outcome Observer assessment severity score; scale between 0 (not itchy at all) and 4 (extremely itchy); the lower the score the better.
Time Frame: MMRM model was used with inputs of the average changes from baseline (BL) to Weeks 1-6, 7-10, 11-14, 15-18, 19-22, 23-26, and other covariates. The average change from BL over Weeks 15-26 is calculated in the model and presented as a single number.
Population: Primary Cohort, defined as participants with genetic testing results consistent with biallelic disease causing variation in ABCB11 (PFIC2, also referred to as BSEP deficiency), based on standard-of-care genotyping, excluding those PFIC2 participants predicted to have complete absence of BSEP function (PFIC2 participants with heterozygosis, biliary diversion, having low or fluctuating sBA levels).
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Groups:
- Primary Cohort Maralixibat: Participants received Maralixibat oral solution (up to 600 microgram per kilogram [mcg/kg]) orally twice daily for 26 weeks.
  Maralixibat: Maralixibat oral solution (up to 600 mcg/kg) orally twice daily for 26 weeks.
- Primary Cohort Placebo: Participants received placebo matched to maralixibat oral solution twice daily for 26 weeks.
  Placebo: Placebo matching to maralixibat orally twice daily for 26 weeks.
Arm/Group | Primary Cohort Maralixibat | Primary Cohort Placebo
Number analyzed (Participants) | 14 | 17
Score on a scale | -1.718 [-2.272 to -1.163] | -0.628 [-1.136 to -0.121]
Statistical Analysis 1: Comparison: Primary Cohort Maralixibat vs Primary Cohort Placebo; The difference between maralixibat and placebo treatment groups in the mean change in the average ItchRO(Obs) severity score between baseline and Weeks 15-26; Test type: Superiority; p = 0.0063, Mixed Models Analysis; Least-Square mean = -1.089, 95% CI 2-sided [-1.845 to -0.334], Standard Error of Mean 0.3691

2. Secondary Outcome: Mean Change in Total sBA Level in the Primary Cohort.
Description: Mean change in total sBA level between baseline and average of Weeks 18, 22 and 26.
Time Frame: Baseline and average of Weeks 18, 22 and 26
Population: Primary Cohort, defined as participants with genetic testing results consistent with biallelic disease causing variation in ABCB11 (PFIC2, also referred to as BSEP deficiency), based on standard-of-care genotyping, excluding those PFIC2 participants predicted to have complete absence of BSEP function (PFIC2 participants with heterozygosis, biliary diversion, having low or fluctuating sBA levels). Two maralixibat participants did not have baseline sBA values and were not included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: μmol/L
Arm/Group | Primary Cohort Maralixibat | Primary Cohort Placebo
Number analyzed (Participants) | 12 | 17
μmol/L | -175.536 [-256.716 to -94.356] | 11.187 [-58.073 to 80.446]
Statistical Analysis 1: Comparison: Primary Cohort Maralixibat vs Primary Cohort Placebo; Test type: Superiority; p = 0.0013, Mixed Models Analysis; Least-Square mean = -186.723, 95% CI 2-sided [-293.454 to -79.992], Standard Error of Mean 51.9501

3. Secondary Outcome: Mean Change in the Average Morning ItchRO(Obs) Severity Score in Participants With PFIC (PFIC1, Nt-PFIC2, PFIC3, PFIC4 and PFIC6)
Description: Mean change in the average morning ItchRO(Obs) severity score between baseline and Week 15 through Week 26 in participants with PFIC (PFIC1, PFIC2, PFIC3, PFIC4 and PFIC6).
  ItchRo(Obs) Severity Score = Itch Reported Outcome Observer assessment severity score; scale between 0 (not itchy at all) and 4 (extremely itchy); the lower the score the better.
Time Frame: Between Baseline and Week 15 through Week 26
Population: Primary cohort plus PFIC1, PFIC3, PFIC4, PFIC6.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Groups:
- PFIC Cohort Maralixibat: After a screening period of up to 6 weeks, subjects were randomized 1:1 to receive either maralixibat or placebo. The Dose Escalation period (4-6 weeks) followed by a stable dosing period (20-22 weeks) and a 7 days Safety Follow-up period for subjects discontinuing early and for subjects not enrolling into the extension Study MRX-503.
- PFIC Cohort Placebo: Participants received a corresponding placebo
Arm/Group | PFIC Cohort Maralixibat | PFIC Cohort Placebo
Number analyzed (Participants) | 33 | 31
score on a scale | -1.811 [-2.178 to -1.444] | -0.610 [-1.000 to -0.221]
Statistical Analysis 1: Comparison: PFIC Cohort Maralixibat vs PFIC Cohort Placebo; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Least-Square mean = -1.200, 95% CI 2-sided [-1.727 to -0.674], Standard Error of Mean 0.2630

4. Secondary Outcome: Mean Change in Total sBA Level in Participants With PFIC (PFIC1, PFIC2, PFIC3, PFIC4 and PFIC6)
Description: Mean change in total sBA level between baseline and average of Weeks 18, 22, and 26 in participants with PFIC (PFIC1, PFIC2, PFIC3, PFIC4 and PFIC6)
Time Frame: Between Baseline and average of Weeks 18, 22 and 26
Population: Primary cohort plus PFIC1, PFIC3, PFIC4 and PFIC6.
Measure: Least Squares Mean (95% Confidence Interval); unit: μmol/L
Arm/Group | PFIC Cohort Maralixibat | PFIC Cohort Placebo
Number analyzed (Participants) | 33 | 31
μmol/L | -157.489 [-200.276 to -114.703] | 2.913 [-42.320 to 48.146]
Statistical Analysis 1: Comparison: PFIC Cohort Maralixibat vs PFIC Cohort Placebo; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Least-Square mean = -160.403, 95% CI 2-sided [-220.836 to -99.970], Standard Error of Mean 30.1827

5. Secondary Outcome: Proportion of ItchRO(Obs) Responders in the Primary Cohort
Description: Proportion of ItchRO(Obs) responders from Week 15 to Week 26 in participants with PFIC2 using the average value from the three 4-week periods (Weeks 15-18, 19-22 and 23-26). The number in the Subject Analysis Set refers to the number of responders.
  ItchRO responders are defined as a subject having a 4-week average morning ItchRO(Obs) severity change from baseline of ≤-1.0 or an average severity score of ≤1.0.
Time Frame: Week 15 to Week 26 using the average value from the three 4-week periods (Weeks 15-18, 19-22 and 23-26)
Population: as for outcome 1
Measure: Number; unit: Number of responders
Arm/Group | Primary Cohort Maralixibat | Primary Cohort Placebo
Number analyzed (Participants) | 14 | 17
Number of responders | 8 | 4
Statistical Analysis 1: Comparison: Primary Cohort Maralixibat vs Primary Cohort Placebo; Test type: Other; p = 0.0736, Bernard's exact test

6. Secondary Outcome: Proportion of sBA Responders in the Primary Cohort
Description: Proportion of sBA responders from Week 18 to Week 26 in participants with PFIC2, using the average value from Weeks 18, 22 and 26 values. The number in the Subject Analysis Set refers to the number of responders.
  sBA responders are defined as a subject having an average sBA level of <102 umol/L (applies only if baseline sBA level was ≥102 umol/L), OR a ≤-75% average percent change from baseline.
Time Frame: Average value from Weeks 18, 22 and 26
Population: as for outcome 1
Measure: Number; unit: Number of responders
Arm/Group | Primary Cohort Maralixibat | Primary Cohort Placebo
Number analyzed (Participants) | 14 | 17
Number of responders | 5 | 1
Statistical Analysis 1: Comparison: Primary Cohort Maralixibat vs Primary Cohort Placebo; Test type: Superiority; p = 0.0410, Bernard's exact test

7. Secondary Outcome: Proportion of ItchRO(Obs) Responders PFIC (PFIC1, PFIC2, PFIC3, PFIC4 and PFIC6)
Description: Proportion of ItchRO(Obs) responders from Week 15 to Week 26 in participants with PFIC (PFIC1, PFIC2, PFIC3, PFIC4 and PFIC6). The number in the Subject Analysis Set refers to the number of responders.
  ItchRO responders are defined as a subject having a 4-week average morning ItchRO(Obs) severity change from baseline of ≤-1.0 OR an average severity score of ≤1.0.
Time Frame: From Week 15 to Week 26
Population: Primary cohort plus PFIC1, PFIC3, PFIC4 and PFIC6.
Measure: Number; unit: Number of responders
Arm/Group | PFIC Cohort Maralixibat | PFIC Cohort Placebo
Number analyzed (Participants) | 33 | 31
Number of responders | 21 | 8
Statistical Analysis 1: Comparison: PFIC Cohort Maralixibat vs PFIC Cohort Placebo; Test type: Superiority; p = 0.0023, Bernard's exact test

8. Secondary Outcome: Proportion of sBA Responders PFIC (PFIC1, PFIC2, PFIC3, PFIC4 and PFIC6)
Description: Proportion of sBA responders from Week 18 to Week 26 in participants with PFIC (PFIC1, PFIC2, PFIC3, PFIC4 and PFIC6). The number in the Subject Analysis Set refers to the number of responders.
  sBA responders are defined as a subject having an average sBA level of <102 umol/L (applies only if baseline sBA level was ≥102 umol/L), or a ≤-75% average percent change from baseline.
Time Frame: Week 18 to Week 26
Population: Primary cohort plus PFIC1, PFIC3, PFIC4 and PFIC6.
Measure: Number; unit: Number of responders
Arm/Group | PFIC Cohort Maralixibat | PFIC Cohort Placebo
Number analyzed (Participants) | 33 | 31
Number of responders | 15 | 2
Statistical Analysis 1: Comparison: PFIC Cohort Maralixibat vs PFIC Cohort Placebo; Test type: Superiority; p = 0.0004, Bernard's exact test

ADVERSE EVENTS:
Time Frame: Baseline to end of treatment (EOT); where EOT can be up to 26 weeks if participant did not early terminate.
Description: The Study Protocol did not require to collect Adverse Events by dose level.
Groups:
- Maralixibat: All participants who received at least 1 dose of maralixibat
- Placebo: All participants who received at least 1 dose of placebo
Arm/Group | Maralixibat | Placebo
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/46
Serious Adverse Events (participants affected / at risk) | 5/47 | 3/46
Other Adverse Events (participants affected / at risk) | 47/47 | 43/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maralixibat (N=47) | Placebo (N=46)
Accidental exposure to product (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Idiopathic pneumonia syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (4) | 0 (0)
Vitamin K deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maralixibat (N=47) | Placebo (N=46)
Blood bilirubin increased (Investigations) | 7 (7) | 4 (4)
Alanine aminotransferase increased (Investigations) | 6 (7) | 3 (3)
Vitamin E decreased (Investigations) | 4 (4) | 3 (3)
Vitamin D decreased (Investigations) | 4 (4) | 2 (2)
International normalised ratio increased (Investigations) | 1 (1) | 4 (5)
Pyrexia (General disorders) | 17 (19) | 13 (20)
Diarrhoea (Gastrointestinal disorders) | 27 (51) | 9 (16)
Abdominal pain (Gastrointestinal disorders) | 10 (16) | 3 (4)
Vomiting (Gastrointestinal disorders) | 3 (3) | 5 (7)
Abdominal pain upper (Gastrointestinal disorders) | 2 (3) | 4 (4)
Constipation (Gastrointestinal disorders) | 4 (4) | 2 (3)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 5 (5)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 8 (11) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 5 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5) | 8 (10)
Upper respiratory tract infection (Infections and infestations) | 3 (6) | 6 (10)
Influenza (Infections and infestations) | 6 (9) | 2 (2)
Coronavirus infection (Infections and infestations) | 3 (3) | 4 (5)
Nasopharyngitis (Infections and infestations) | 5 (8) | 2 (3)
Gastroenteritis (Infections and infestations) | 3 (4) | 2 (2)
Vitamin D deficiency (Metabolism and nutrition disorders) | 4 (5) | 4 (5)
Vitamin E deficiency (Metabolism and nutrition disorders) | 3 (3) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2022-05-10): https://cdn.clinicaltrials.gov/large-docs/30/NCT03905330/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-29): https://cdn.clinicaltrials.gov/large-docs/30/NCT03905330/SAP_001.pdf